CLINICAL TRIAL: NCT01075061
Title: Study of a Large Family With Congenital Mirror Movements : From Underlying Pathophysiology to Culprit Gene Identification : MOMIC
Brief Title: Study of a Large Family With Congenital Mirror Movements : From Underlying Pathophysiology to Culprit Gene Identification PROJET " MOMIC "
Acronym: MOMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C09-06; 2009-A00490-57 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-02-04; First posted 2010-02-24 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Congenital mirror movement, physiopathology, imaging, transcranial magnetic stimulation, candidate gene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy volunteers (Other): healthy volunteers
  Interventions: Other: healthy volunteers
- Kallmann (Other): Kallmann syndrome patients
  Interventions: Other: Kallmann
- Congenital Mirror Movement (Other): patients with CMM
  Interventions: Other: Congenital Mirror Movement

INTERVENTIONS:
Other: healthy volunteers — morphological and functional brain MRI; transcranial magnetic stimulation
  Arms: healthy volunteers
Other: Kallmann — morphological and functional brain MRI; transcranial magnetic stimulation
  Arms: Kallmann
Other: Congenital Mirror Movement — morphological and functional brain MRI; transcranial magnetic stimulation
  Arms: Congenital Mirror Movement

SUMMARY:
Mirror movements are involuntary, symmetrical and simultaneous movements occurring on one side of the body that accompany controlateral voluntary movements. Congenital mirror movements (CMM) are characterized by childhood onset and the absence of additional manifestations. The aim of this study is to unravel the pathophysiology of the CMM that remains poorly elucidated. The combination of imaging studies and neurophysiological studies using transcranial magnetic stimulation in a homogeneous and relatively large group of patient is likely to allow us to better understand the underlying pathophysiology of the disorder. Using a linkage analysis approach we will try to identify a locus associated with CMM and related candidate genes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 11 to 82 years
* Members of the family of interest displaying mirror movements or being obligatory asymptomatic carrier, without additional manifestation or malformation; or patient with genetically proven Kallmann syndrome and mirror movements.
* No contraindication for MRI or TMS study

Exclusion Criteria:

* inability to provide an informed consent
* Simultaneous participation in another clinical trial
* Treatment that modulate cortical excitability (for the TMS part of the study only)

Ages: 11 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
- To unravel the pathophysiology of congenital mirror movements - To identify a locus and candidate genes associated with CMM | 08/2011

SECONDARY OUTCOMES:
- To study patients with Kallmann syndrome and associated MM based on the same methods and hypothesis | 08/2011

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel ROZE, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Fédération des Maladies du Système Nerveux, Hôpital Pitié Salpétrière, Paris, France

REFERENCES:
- [Background] Depienne C, Cincotta M, Billot S, Bouteiller D, Groppa S, Brochard V, Flamand C, Hubsch C, Meunier S, Giovannelli F, Klebe S, Corvol JC, Vidailhet M, Brice A, Roze E. A novel DCC mutation and genetic heterogeneity in congenital mirror movements. Neurology. 2011 Jan 18;76(3):260-4. doi: 10.1212/WNL.0b013e318207b1e0. PMID 21242494